CLINICAL TRIAL: NCT03643640
Title: Evaluation of a Web-based Psychological Intervention as add-on to Care as Usual in Breast Cancer Survivors: Effect on Lifestyle and Psychometric Outcome
Brief Title: Evaluating a Novel Web-based Intervention for Breast Cancer Survivors
Acronym: OPTIMUNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Dortmund (Other)
Collaborators: University of Leipzig (Other); Gaia AG (Industry)
Responsible Party: Principal Investigator, Carsten Watzl, Scientific Director, IfADo, Technical University of Dortmund
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Optimune Trial Add-on
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimune (Experimental): Optimune is an web-based psychological intervention for women with breast cancer. Beyond established CBT techniques targeting depression, anxiety, and fatigue, this intervention specifically includes elements that have shown effects on markers of immune status and inflammation, including sleep, stress management (e.g., mindfulness-based techniques) and lifestyle optimization (dietary and physical activity advice). Content is continuously adapted to users' concerns and needs. It contains interactive dialogues that can be accessed via computer or smart-phone, illustrations, audio files and motivating text messages. Optional daily text messages with motivational content accompany the program. The program can be accessed for 365 days after registration.
  Interventions: Behavioral: Optimune
- Care-as-Usual (Active Comparator): As in the experimental arm, participants are free to continue to engage with any treatment they require (i.e., CAU). However, they will receive access to Optimune six months post-baseline (i.e., wait list with respect to Optimune access).
  Interventions: Other: Care-As-Usual

INTERVENTIONS:
Behavioral: Optimune — Optimune is a web-based psychological intervention developed for women with breast cancer.
  Arms: Optimune
Other: Care-As-Usual — Participants are free to continue to engage with any treatment they require (i.e., CAU).
  Arms: Care-as-Usual

SUMMARY:
The trial aims to evaluate the effectiveness of a novel web-based intervention (Optimune), which was designed to introduce relevant cognitive-behavioral therapy (CBT) techniques to women with breast cancer who are past the active eradication phase. The present study will test the hypothesis that Optimune has an impact on lifestyle parameters and psychometric outcomes. Therefore, 360 woman with breast cancer will be recruited and randomized to two groups: (1) a control group, in which they may engage with any treatment (Care-as-Usual, CAU) and receive access to Optimune after a delay of 3 months (i.e., CAU/wait list control group), or (2) to a treatment group that immediately receives 12-month access to Optimune and may also use CAU. The primary outcome measure is the effect on quality of life, physical activity and diet three month post-baseline.

DETAILED DESCRIPTION:
Depression and fatigue is common in breast cancer survivors and its presence is associated with personal suffering, increased inflammatory activity, and worse prognosis. While in the phase of acute treatment many women receive short-term psychological support to better cope with the situation, this is not standard of care in the years following. Web-based psychological interventions are easily accessible and preliminary evidence suggests that such interventions can be effective. However, no trial has yet examined whether a CBT-based internet intervention designed to meet the needs of breast cancer survivors can achieve effects on lifestyle parameters and psychometric outcomes, when offered as adjunct to care as usual.

In this study, the investigators will investigate treatment effects of the novel web-based program Optimune when added to treatment as usual. Beyond established CBT techniques targeting depression, anxiety, and fatigue, this intervention specifically includes elements that have shown effects on markers of immune status and inflammation, including sleep and stress management (e.g., mindfulness-based techniques) and lifestyle optimization (dietary and physical activity advice). The delivery and training of content is continuously individualized to match users' preferences and needs, based on responses within the program. The intervention is delivered via the internet and protected by individually assigned passwords. The program can be accessed for 365 days after registration.

This randomized controlled trial will include 360 women with breast cancer who are past the active eradication phase. Participants will be recruited from various settings, including web-based advertisement and internet forums/groups. Participants will be randomly assigned to either (1) a control group, in which they receive care as usual (CAU) and are given access to the web-based intervention (Optimune) after a delay of 3 months (i.e., CAU/wait list control group), or (2) a treatment group that may also use CAU and in addition immediately receives 12-month access to the web-based intervention (Optimune). Measurements are collected at pre-treatment (T0) three months (T1) and six months (T2).

ELIGIBILITY:
Eligible are women who

* had breast cancer diagnosed less than 5 years ago
* completed acute treatment for breast cancer at least 1 month ago. This applies for surgery, chemotherapy or radiation, whichever occurred last. (Prophylactic treatment with anti-hormones like tamoxifene, aromatase-inhibitors or bisphosphonates is allowed).
* are competent in German language
* provide written consent to study procedures
* are willing to provide the discharge letter from oncology (to verify diagnosis and therapies)

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Determination of Quality of Life using the WHOQOL-BREF | Change from baseline to 3 months (also assessed at 6 months post-baseline)
  Quality of Life will be measured using the World Health Organization Quality of Life Questionnaire (WHOQOL-BREF), which is a shorter version of the original instrument. Scale Range: 26 to 130.
  The WHOQOL-BREF is a 26-item, 5-point rating scale. It measures the following broad domains: physical health, psychological health, social relationships, and environment. Response options range from 1, indicating "very dissatisfied" to 5, indicating "very satisfied" and relate to the last two weeks.
  Higher scores on the WHOQOL-BREF correspond to higher self-reported levels of quality of life.
Determination of Physical Activity using the International Physical Activity Questionnaire | Change from baseline to 3 months (also assessed at 6 months post-baseline)
  Physical Activity will be measured using the short version of the International Physical Activity Questionnaire (IPAQ - short).
  The short version of the IPAQ is a 7-item questionnaire that assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives. Open-ended questions surrounding individuals' last 7-day recall of physical activity are considered to estimate total physical activity min/week and time spent sitting.
  Interpretation: Three levels (categories) of physical activity are proposed: low, moderate and high.
Determination of Diet Quality using the Food Quality Questionnaire | Change from baseline to 3 months (also assessed at 6 months post-baseline)
  Diet Quality will be measured using the Food Quality Questionnaire (FQQ). Scale Range: 0 to 39.
  The FQQ is a 10-item, 5-point rating scale. The FQQ is a short food frequency questionnaire, which includes 10 food items on a 5-point rating scale. It focuses on fruit, vegetables, high-sugar foods, processed food, meat and drinks. The aim of the tool is to measure diet quality. Response options range from 0, indicating "daily" to 3" indicating, "once or never". Interpretation: A global diet quality score can be obtained by averaging all the items on the FQQ.

SECONDARY OUTCOMES:
Determination of cancer-related fatigue using the Brief Fatigue Inventory Questionnaire | Change from baseline to 3 months (also assessed at 6 months post-baseline)
  Fatigue will be measured using the Brief Fatigue Inventory Questionnaire (BFI-9) questionnaire. Scale Range: 0 to 90.
  The BFI is a 9-item, 11-point rating scale. The first three questions measure fatigue severity from 0, indicating "no fatigue," to 10, indicating "as bad as you can imagine," at current, usual, and worst levels. The following six questions assess fatigue interference with daily activities. Response options range from 0, indicating "does not interfere," to 10, indicating, "completely interferes." Interpretation: A global fatigue score can be obtained by averaging all the items on the BFI.
  Higher scores on the BFI correspond to greater self-reported levels of fatigue
Determination of cancer-related emotional stress | Change from baseline to 3 months (also assessed at 6, 9 and 12 months post-baseline)
  Cancer-related emotional stress will be measured using the standardized IES-R (Impact of Event Scale) Questionnaire. Scale Range: 0 to 88 The IES-R is a 22-item self-report measure that assesses subjective distress caused by traumatic events. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score (ranging from 0 to 88) and subscale scores can also be calculated for the Intrusion, Avoidance, and Hyperarousal subscales.
  Interpretation: Higher scores correspond to greater self-reported levels of post-traumatic stress.
Determination of depression | Change from baseline to 3 months (also assessed at 6 months post-baseline)
  Depression will be measured using the standardized PHQ-9 (Patient Health Questionnaire). Scale Range: 0 to 27 The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression.
  Interpretation: Higher scores correspond to greater self-reported levels of depression.
Determination of anxiety | Change from baseline to 3 months (also assessed at 6 months post-baseline)
  Anxiety will be measured using the standardized GAD-7 (Generalized Anxiety Disorder) questionnaire. Scale Range: 0 to 21 The GAD-7 is an instrument for screening, diagnosing, monitoring and measuring the severity of anxiety. GAD-7 scores of 5, 10, and 15 represents mild, moderate, and severe anxiety.
  Interpretation: Higher scores correspond to greater self-reported levels of anxiety.
Determination of fear of progression | Change from baseline to 3 months (also assessed at 6 months post-baseline)
  Fear of progression will be measured using the standardized PA-F12 (Fear of progression) questionnaire. Scale Range: 12 - 60 The PAF-12 items are scored on a five-point Likert Scale ranging from 1 ('never') to 5 ('very often'), higher values indicating higher levels of anxiety.
  Interpretation: Higher scores correspond to greater self-reported levels of fear of progression.
Determination of insomnia | Change from baseline to 3 months (also assessed at 6 months post-baseline)
  Insomnia will be measured using the standardized - ISI (Insomnia Severity Index), Scale Range: 0 - 28, higher values indicating increasing severity of insomnia
Determination of usefulness of the program | Assessed at 3 and 6 months
  Usefulness of the program will be measured by a questionnaire
Determination of Negative Effects | Assessed at 3 and 6 months
  Negative Effects will be measured using the standardized INEP (Inventory for the Assessment of Negative Effects of Psychotherapy) questionnaire.

OTHER OUTCOMES:
Determination of recurrence of breast cancer (local relapse or remote metastasis) | Change from baseline to 3 months (also assessed at 6 months post-baseline)
  Recurrence of breast cancer (local relapse or remote metastasis) will be determined by a questionnaire
Frequency of common cold or virus flu | Change from baseline to 3 months (also assessed at 6 months post-baseline)
  Frequency of common cold or virus flu will be determined by a questionnaire
Frequency of unscheduled medical encounters | Change from baseline to 3 months (also assessed at 6 months post-baseline)
  Frequency of unscheduled medical encounters will be determined by a questionnaire
Body Mass Index | Change from baseline to 3 months (also assessed at 6 months post-baseline)
  Height and weight will be determined by a questionnaire
Psychotherapy | Change from baseline to 3 months (also assessed at 6 months post-baseline)
  A questionnaire will determine if a psychotherapy has started during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Watzl, PhD, Principal Investigator — Leibniz Research Center (IfADo), TU Dortmund
Locations (2):
- Germany (2):
  - Technical University of Dortmund, Leibniz Research Centre for Working Environment and Human Factors, Dortmund
  - University Medical Center Leipzig, Department of Medical Psychology and Medical Sociology, Section Psychosocial Oncology, Leipzig

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data shall be made available upon request for projects such as meta-analyses after completion of the study
Time Frame: after completion of the study
Access Criteria: available upon request

REFERENCES:
- [Derived] Holtdirk F, Mehnert A, Weiss M, Mayer J, Meyer B, Brode P, Claus M, Watzl C. Results of the Optimune trial: A randomized controlled trial evaluating a novel Internet intervention for breast cancer survivors. PLoS One. 2021 May 7;16(5):e0251276. doi: 10.1371/journal.pone.0251276. eCollection 2021. PMID 33961667
- [Derived] Holtdirk F, Mehnert A, Weiss M, Meyer B, Watzl C. Protocol for the Optimune trial: a randomized controlled trial evaluating a novel Internet intervention for breast cancer survivors. Trials. 2020 Jan 29;21(1):117. doi: 10.1186/s13063-019-3987-y. PMID 31996235